CLINICAL TRIAL: NCT04603339
Title: ReStOre@Home: Feasibility Study of a 12-week Multidisciplinary Telehealth Rehabilitation Programme for Survivors of Upper Gastrointestinal (UGI) Cancer
Acronym: ReStOre@Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Prof Juliette Hussey, Professor of Physiotherapy, University of Dublin, Trinity College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIFA-2018-009 - ReStOre@Home
Record Dates: First submitted 2020-09-21; First posted 2020-10-26 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Oesophageal Cancer; Gastric Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Single arm trial, all participants will receive the intervention
  Interventions: Other: Multidisciplinary rehabilitation programme delivered via telehealth

INTERVENTIONS:
Other: Multidisciplinary rehabilitation programme delivered via telehealth — 12 week programme of;
  1) Physiotherapy led aerobic and resistance exercise 2)1:1 Dietetics Counselling 3) Group Multidisciplinary Education Sessions

SUMMARY:
Feasibility study of a 12-week multidisciplinary telehealth rehabilitation programme for survivors of upper gastrointestinal (UGI) cancer

DETAILED DESCRIPTION:
A single arm feasibility study will be conducted to examine the feasibility of delivering the 12-week ReStOre programme (aerobic and resistance physiotherapy led-exercise, 1:1 dietary counselling and group education sessions) via telehealth to a cohort of upper gastrointestinal cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* be ≥ three months post oesophagectomy, total gastrectomy
* ± neo-adjuvant/adjuvant chemo/chemoradiotherapy with curative intent
* adjuvant therapy must be completed
* access to home broadband

Exclusion Criteria:

* Ongoing serious post-operative morbidity
* Evidence of active or recurrent disease.

In addition those with any serious co-morbidity that would impact on exercise participation will be excluded including those with;

* Uncontrolled hypertension (resting systolic blood pressure >180mmHg and/or diastolic >100mmHg)
* Recent serious cardiovascular events (within 12 months) including, but not limited to cerebrovascular accident, and myocardial infarction
* Unstable cardiac, renal, lung, liver or other severe chronic disease
* Uncontrolled atrial fibrillation
* Left ventricular function <50%.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Feasibility - Recruitment | Through study completion approx 1 year
  Feasibility will be determined by recruitment rate, the number of eligible participants who consent to participation.
Feasibility - adherence | From baseline (T0) to immediately after the program intervention (T1)
  Feasibility will also be determined by adherence to the trial intervention, the number of prescribed intervention sessions completed.
Feasibility - acceptability of the intervention (1) | Immediately after the program intervention (T1)
  Feasibility will also be determined by the acceptability of the programme. Acceptability of the telehealth programme will be assessed by the Telehealth Usability Questionnaire (TUQ).
  The Telehealth Usability scale is a 5 point likert scale where 1 = completely disagree, and 5 =fully agree, Higher ratings indicate better usability.
Feasibility - acceptability of the intervention (2) | Duration of the trial i.e. From enrolment of the first participant until completion of the final participants post-intervention assessment (Time period of up to 12 months).
  Acceptability of the intervention will be further determined by a qualitative approach.Interviews will be carried out with participants post-intervention to gain their perspectives of the impact of the program on physical and mental well-being and the suitability of the programme to delivery via telehealth

SECONDARY OUTCOMES:
Change in Cardiorespiratory Fitness from Baseline | Baseline (T0), Immediately after the program intervention (T1)
  Cardiorespiratory fitness will be determined by Cardiopulmonary Exercise Test (CPET)
Physical Performance | Baseline (T0), Immediately after the program intervention (T1)
  Physical Performance will be measured with the Short Physical Performance Battery
Hand Grip Strength | Baseline (T0), Immediately after the program intervention (T1)
  Hand Grip strength will be measured with hand held dynamometry
Physical Activity | Baseline (T0), Immediately after the program intervention (T1)
  Physical activity will be measured using the Godin Shepherd Leisure-Time Exercise Questionnaire. A score of 24 indicates the individual is active, 14-23 indicates moderately active, and less than 14 indicates sedentary/ insufficiently active.
Weight | Baseline (T0), Immediately after the program intervention (T1)
  Weight will be recorded by standard measures and reported in kilograms (kg).
Height | Baseline (T0), Immediately after the program intervention (T1)
  Height will be recorded by standard measures and reported in meters (m)
Body Mass Index | Baseline (T0), Immediately after the program intervention (T1)
  Body Mass Index (BMI) will be calculated as weight (kg)/height (meters(m2)) and reported in kilograms/metres squared (kg/m2).
Circumferential Measurements | Baseline (T0), Immediately after the program intervention (T1)
  Mid-arm circumference and waist circumference will be measured with a flexible tape measure and reported in centimeters (cm)
Health Related Quality of Life measured by the European Organisation for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30) | Baseline (T0), Immediately after the program intervention (T1)
  Quality of Life will be determined by the European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30).
  Scores are reported on a linear scale from 0-100. A high score in a functional scale indicates greater function. A high score in a symptom scale indicates greater symptom burden.
Oesophago-gastric cancer specific Health Related Quality of Life will measured by the European Organisation for the Research and Treatment of Cancer Oesophago-gastric Cancer Subscale the EORTC-QLQ-OG25. | Baseline (T0), Immediately after the program intervention (T1)
  Oesophagogastric cancer specific quality of life will be determined by the EORTC-QLQ-OG25 subscale.
  Scores are reported on a linear scale from 0-100. A high score in a functional scale indicates greater function. A high score in a symptom scale indicates greater symptom burden.
Fatigue | Baseline (T0), Immediately after the program intervention (T1)
  Fatigue will be assessed using the Multidimensional Fatigue Inventory (MFI-20) questionnaire. It is scored from 0-20. A cut off score of >or =13 indicates severe fatigue.
Bio-sample Collection | Baseline (T0), Immediately after the program intervention (T1)
  Serum, Plasma and Whole Blood samples will be collected at each time-point to establish a survivorship Biobank for UGI cancer. These samples will be stored in the biobank for future to be determined studies.

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Hussey, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Trinity College Dublin, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Neill L, Guinan E, Brennan L, Doyle SL, O'Connor L, Sheill G, Smyth E, Fairman CM, Segurado R, Connolly D, O'Sullivan J, Reynolds JV, Hussey J. ReStOre@Home: Feasibility study of a virtually delivered 12-week multidisciplinary rehabilitation programme for survivors of upper gastrointestinal (UGI) cancer - study protocol. HRB Open Res. 2021 May 4;3:86. doi: 10.12688/hrbopenres.13185.2. eCollection 2020. PMID 34046552